CLINICAL TRIAL: NCT03506633
Title: Impacts of Mitochondrial-targeted Antioxidant on Leg Function, Leg Blood Flow and Skeletal Muscle Mitochondrial Function in Peripheral Artery Disease Patients
Brief Title: Impacts of Mitochondrial-targeted Antioxidant on Peripheral Artery Disease Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 0086-18-FB
Record Dates: First submitted 2018-04-13; First posted 2018-04-24 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Peripheral Arterial Disease; Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — mitoquinone

STUDY DESIGN:
Intervention Model Description: 1:1 Randomized, cross-over, double-blinded design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MitoQ-Placebo (Experimental): Participants will be tested on two different days, first day will be baseline and MitoQ and second day will be Placebo. Testing will take place forty-minutes after MitoQ/placebo intake. There will be a 2-week washout between testing days.
  Interventions: Dietary Supplement: MitoQ
- Placebo-MitoQ (Experimental): Participants will be tested on two different days, first day will be baseline and Placebo and second day will be MitoQ. Testing will take place forty-minutes after placebo/MitoQ intake. There will be a 2-week washout between testing days.
  Interventions: Dietary Supplement: MitoQ

INTERVENTIONS:
Dietary Supplement: MitoQ — A mitochondrial-targeting antioxidant "MitoQ" or a placebo will be given to each participant in a crossover, double-blinded design and measures of leg function and leg blood flow will be measured.

SUMMARY:
Peripheral artery disease (PAD) is a common cardiovascular disease, in which narrowed arteries reduce blood flow to the limbs, causing pain, immobility and in some cases amputation or death. PAD patients have shown higher levels of systemic and skeletal muscle inflammation due to the impaired oxygen transfer capacity of these blood vessels. This attenuated oxygen transfer capacity causes hypoxic conditions in the skeletal muscle and results in mitochondrial dysfunction and elevated reactive oxygen species (ROS). These harmful byproducts of cell metabolism are the major cause of intermittent claudication, defined as pain in the legs that results in significant functional limitations. One potential defensive mechanism to these negative consequences may be having higher antioxidant capacity, which would improve blood vessel vasodilatory function, enabling more blood to transfer to the skeletal muscles. Therefore, the purpose of this project is to examine the impact of mitochondrial targeted antioxidant (MitoQ) intake on oxygen transfer capacity of blood vessels, skeletal muscle mitochondrial function, leg function, and claudication in participants with PAD. Blood vessel oxygen transfer capacity in the leg will be assessed in the femoral and popliteal arteries. Skeletal muscle mitochondrial function and ROS levels will be analyzed in human skeletal muscle via near infrared spectroscopy and through blood samples. Leg function will be assessed by walking on a force platform embedded treadmill and claudication times will be assessed with the Gardner maximal walking distance treadmill test.

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a common cardiovascular disease, in which narrowed arteries reduce blood flow to the limbs, causing pain, immobility and in some cases amputation or death. Previous studies reported that atherosclerotic lesions are distributed non-uniformly in the leg arteries, and the resulting impaired blood flow, and concomitant reduced oxygen delivery to skeletal muscle results in the pathophysiology of PAD. PAD patients have shown higher levels of systemic and skeletal muscle inflammation due to the impaired oxygen transfer capacity of these blood vessels. This attenuated oxygen transfer capacity causes hypoxic conditions in the skeletal muscle and results in mitochondrial dysfunction and elevated reactive oxygen species (ROS). These harmful byproducts of cell metabolism are the major cause of intermittent claudication, defined as pain in the legs that results in significant functional limitations.

One potential defensive mechanism to these negative consequences may be having higher antioxidant capacity, which would improve blood vessel vasodilatory function, enabling more blood to transfer to the skeletal muscles. MitoQ, a derivative of CoQ10, is a commercial antioxidant that counteracts this oxidative stress within the mitochondria. High ROS levels have been positively correlated with reduced Nitric oxide (NO) bioavailability, which limits the ability of the blood vessels to dilate, thereby increasing the occlusion that leads to claudication in PAD patients. MitoQ should reduce these ROS levels and increase vasodilatory function. However, the influence of MitoQ intake on leg blood flow, ROS production, claudication and leg function has not yet been investigated in this disease population.

Therefore, the purpose of this project is to examine the impact of mitochondrial targeted antioxidant (MitoQ) intake on oxygen transfer capacity of blood vessels, skeletal muscle mitochondrial function, leg function, and claudication in participants with PAD. Blood vessel oxygen transfer capacity in the leg will be assessed in the femoral and popliteal arteries. Skeletal muscle mitochondrial function and ROS levels will be analyzed in human skeletal muscle via near infrared spectroscopy and through blood samples. Leg function will be assessed by walking on a force platform embedded treadmill and claudication times will be assessed with the Gardner maximal walking distance treadmill test.

ELIGIBILITY:
Inclusion Criteria:

* Able to give written, informed consent
* Demonstrated positive history of chronic claudication
* History of exercise limiting claudication
* Ankle/brachial index < 0.90 at rest
* Stable blood pressure regimen, stable lipid regimen, stable diabetes regimen and risk factor control for 6 weeks prior to study entry
* 50-85 years old

Exclusion Criteria:

* Resting pain or tissue loss due to Peripheral artery disease (PAD), Fontaine stage III and IV
* Acute lower extremity ischemic event secondary to thromboembolic disease or acute trauma
* Walking capacity limited by conditions other than claudication including leg (joint/musculoskeletal, neurologic) and systemic (heart, lung disease) pathology

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2022-01-17 (Actual); Study Completion 2022-01-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Song-Young Park, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska - Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MitoQ-Placebo: Subjects will be tested on two different days, first day will be baseline and MitoQ and second day will be Placebo. Testing will take place forty-minutes after MitoQ/placebo intake. There will be a 2-week washout between testing days.
  MitoQ: A mitochondrial-targeting antioxidant "MitoQ" or a placebo will be given to each subject in a crossover, double-blinded design and measures of leg function and leg blood flow will be measured.
- Placebo-MitoQ: Subjects will be tested on two different days, first day will be baseline and Placebo and second day will be MitoQ. Testing will take place forty-minutes after placebo/MitoQ intake. There will be a 2-week washout between testing days.
  MitoQ: A mitochondrial-targeting antioxidant "MitoQ" or a placebo will be given to each subject in a crossover, double-blinded design and measures of leg function and leg blood flow will be measured.
Period: First Intervention (1 Day)
Arm/Group | MitoQ-Placebo | Placebo-MitoQ
Started | 8 | 6
Completed | 8 | 6
Not Completed | 0 | 0
Period: Washout (14 Days)
Arm/Group | MitoQ-Placebo | Placebo-MitoQ
Started | 8 | 6
Completed | 7 | 6
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention (1 Day)
Arm/Group | MitoQ-Placebo | Placebo-MitoQ
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 13 patients with peripheral artery disease were recruited to participate in this randomized crossover study design
Groups:
- Total: Total of all reporting groups
Arm/Group | MitoQ-Placebo | Placebo-MitoQ | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 5 | 4 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (8.4) | 71.5 (8.4) | 71.5 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 3 | 3 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 6 | 6 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Endothelial Function
Description: Flow-mediated dilation will be used to measure vasodilation in the brachial artery, and blood flow in the femoral and popliteal arteries. This is measured in percents. Scale range is approximately 8-12% for healthy populations. A higher value represents a better outcome.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: % dilation
Groups:
- MitoQ: Subjects will be tested on two different days, first day will be baseline and MitoQ and second day will be Placebo. Testing will take place forty-minutes after MitoQ/placebo intake. There will be a 2-week washout between testing days.
  MitoQ: A mitochondrial-targeting antioxidant "MitoQ" or a placebo will be given to each subject in a crossover, double-blinded design and measures of leg function and leg blood flow will be measured.
- Placebo: Subjects will be tested on two different days, first day will be baseline and Placebo and second day will be MitoQ. Testing will take place forty-minutes after placebo/MitoQ intake. There will be a 2-week washout between testing days.
  MitoQ: A mitochondrial-targeting antioxidant "MitoQ" or a placebo will be given to each subject in a crossover, double-blinded design and measures of leg function and leg blood flow will be measured.
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 13 | 13
% dilation | 6.13 (2.1) | 3.78 (1.13)

2. Secondary Outcome: Walking Function
Description: Subject will walk on a treadmill starting at a speed of 2.0 mph for two minutes with 0% incline. Every two minutes the treadmill incline will increase by 2% up to a maximum of 14%. The subject will be asked to walk until they feel pain in there legs, at which point the test will stop. This is measured in meters (distance) and seconds (time). Scale range is ~800 meters and 840 for healthy populations. A higher value represents a better outcome. This assessment occurred on two separate days (one for each intervention).
Time Frame: 2 days (1 day for MitoQ and 1 day for Placebo)
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 13 | 13
meters | 451.07 (217.14) | 404.49 (218.09)

3. Secondary Outcome: Oxidative Stress
Description: Blood draws will be taken to measure oxidative stress markers in the blood. This is measured in units per milliliter (U/mL). Measures of oxidative stress are approximately 70-80 U/mL in healthy populations. A lower value represents a better outcome.
Time Frame: 2 days
Measure: Mean (Standard Error); unit: U/mL
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 13 | 13
U/mL | 29.55 (1.62) | 34.14 (0.98)

4. Secondary Outcome: Skeletal Muscle Oxygenation
Description: Near-infrared spectroscopy will be used to measure leg muscle oxygenation. Measures of oxygenation are measured in percents. Scale range is ~70-90% in healthy populations. A higher value represents a better outcome.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: percentage of oxygenation
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 13 | 13
percentage of oxygenation | 48.1 (19.3) | 30.7 (18.2)

5. Secondary Outcome: Autonomic Nervous System Activity
Description: Autonomic nervous system function will be measured non-invasively using heart rate variability via the head-up tilt test. Raw R-R interval data will be converted to time frequency domain with the wavelet transform across the frequency intervals 0.04-0.15 Hz (low-frequency, (LF)) and 0.15-0.4 Hz (high-frequency, HF). Units for both will be expressed as ms^2. Final outcome measure will be the ratio of LF/HF, which is a unitless ratio to indicate sympathetic-to-parasympathetic nervous system function.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 13 | 13
ratio | 3.6 (2.3) | 2.7 (1.8)

6. Secondary Outcome: Microvascular Function
Description: Microvascular function will be assessed using near-infrared spectroscopy. NIRS measurements were taken continuously throughout the entire protocol at a sampling rate of 10 Hz. Hemoglobin and myoglobin possess indistinguishable spectral characteristics in the NIRS signal; therefore, the signal is considered to be primarily derived from Hb. The signals were analyzed according to a modified Beer- Lambert's law, and a constant differential path length factor was not used due to the assumption that constant optical scattering of the photons has been demonstrated to affect alterations in NIRS signals. Data were expressed as relative changes with respect to baseline as a percentage (TOI). Tissue reoxygenation was estimated by calculating the initial slope of TOI recovery, which has been used as an index of microvascular function.
Time Frame: 2 days
Measure: Mean (Standard Deviation); unit: % reoxygenation rate
Arm/Group | MitoQ | Placebo
Number analyzed (Participants) | 13 | 13
% reoxygenation rate | 48.1 (18.8) | 32.3 (17.9)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | MitoQ | Placebo
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/33/NCT03506633/Prot_SAP_001.pdf